CLINICAL TRIAL: NCT05955729
Title: Effect of a Short Nap During the Night Shift of Healthcare Workers on Endothelial Function: NAP-WORK Randomized Controlled Study
Brief Title: Effect of a Short Nap During the Night Shift of Healthcare Workers on Endothelial Function
Acronym: NAP-WORK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23CH138; 2023-A01109-36 (Other: ANSM)
Record Dates: First submitted 2023-06-23; First posted 2023-07-21 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volonteers
Keywords: Nap; Endothelial function; Shift work; Nurses
MeSH Terms: interventions — RE1-silencing transcription factor; Electrocardiography, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nap group (Experimental): The experimental group will be allocated to do a 30-min on-duty nap during night work, in a dedicated room between 1 am and 4 am.
  Interventions: Behavioral: On-duty Nap; Device: EndoPAT; Device: Popmeter®; Device: Panasonic EW3109; Device: ECG Holter; Biological: Fasting blood sample; Other: Pichot fatigue scale; Other: French version of the Recovery Needs Scale (BRD); Other: The Short-Form 36 (SF-36); Other: Pittsburgh Sleep Quality Index (PSQI); Other: Epworth questionnaire; Other: The Karolinska Sleepiness Scale; Device: Actimeter
- Control group (Active Comparator): The control group will be allocated to rest in a dedicated room without napping between 1 am and 4 am.
  Interventions: Behavioral: Control condition (30-min rest); Device: EndoPAT; Device: Popmeter®; Device: Panasonic EW3109; Device: ECG Holter; Biological: Fasting blood sample; Other: Pichot fatigue scale; Other: French version of the Recovery Needs Scale (BRD); Other: The Short-Form 36 (SF-36); Other: Pittsburgh Sleep Quality Index (PSQI); Other: Epworth questionnaire; Other: The Karolinska Sleepiness Scale; Device: Actimeter

INTERVENTIONS:
Behavioral: On-duty Nap — For 12 weeks, an opportunity for a 30-minute nap during the night shift, between 1 a.m. and 4 a.m., in a quiet room with facilities for lying down.
  Arms: Nap group
Behavioral: Control condition (30-min rest) — For 12 weeks, an opportunity for a 30-minute rest during the night shift, between 1 a.m. and 4 a.m., in a quiet room without facilities for lying down or napping.
  Arms: Control group
Device: EndoPAT — The EndoPAT device® measures vascular reactivity after a 5-minute occlusion on one arm.
  This device measures changes in vascular tone induced by the endothelium at fingertip level using a pair of plethysmographic sensors. The measurement consists of performing a reference recording for 5 minutes on the 2 arms, then a test arm is chosen to perform an occlusion for 5 minutes while continuing the recording.
Device: Popmeter® — The tool is connected to the caregiver's finger and toe via photodiode sensors. Its simple operation enables reproducible measurement of the propagation speed of the pulse wave in 14 seconds.
Device: Panasonic EW3109 — Diastolic and systolic blood pressure measured 3 times in succession using an automatic blood pressure monitor (Panasonic EW3109) in the sitting position on the left arm.
  Other Names: automatic blood pressure device
Device: ECG Holter — The Holter takes an ECG during the subject's daily activities at home.
  Other Names: portable electrocardiogram
Biological: Fasting blood sample — 15 ml blood sample (venous sampling) will be taken to measure inflammatory biomarkers (hsCRP, IL-6 TNF-α, IL-1β) and blood markers of endothelial function (NO, CRP, SOD, IL-18).
Other: Pichot fatigue scale — The Pichot fatigue scale is an 8-item questionnaire, with a score above 22 indicating excessive fatigue.
Other: French version of the Recovery Needs Scale (BRD) — BRD questionnaire consists of 11 items coded 0 or 1. A score is calculated for each participant, multiplied by 10 to give a score ranging from 0 to 100. The greater the need for recovery, the higher the score.
Other: The Short-Form 36 (SF-36) — The SF-36 questionnaire is used to assess quality of life. It comprises 8 sub-scores ranging from 0 (minimum quality of life) to 100 (maximum well-being).
Other: Pittsburgh Sleep Quality Index (PSQI) — 24-question sleep quality assessment scale, a score > 5 indicates poor sleep quality
Other: Epworth questionnaire — 8-question sleepiness assessment scale, a score above 10 indicates excessive sleepiness
Other: The Karolinska Sleepiness Scale — The Karolinska Sleepiness Scale measures daytime sleepiness on a 9-point scale, based on 5 states and 4 intermediate states that are not verbally indicated.
Device: Actimeter — An actimeter will be worn on the non-dominant wrist, uninterrupted day and night, for 7 consecutive days.

SUMMARY:
Night shift work is well known to cause health disruption in short and long term. It has been reported that among healthcare workers, nurses slept less than 6 h/24h. Consequences of such short sleep duration has been associated to long term issues such as endothelial dysfunction associated with cardiovascular diseases, arterial hypertension and type 2 diabetes. Countermeasures such as nap at work has potential effects on reducing the prevalence of cardiovascular diseases. However, to our knowledge, no studies have objectively investigated the effects of napping on endothelial function in a longitudinal design. Therefore, this study aims to investigate the effect of a 30 minutes on-duty nap during night work for 12 weeks on caregivers endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Being a paramedical caregiverr (nurse or care assistant) at Saint-Etienne University Hospital
* Be aAged between 18 and 65
* Working at least 80% of a full-time equivalent post
* Working 12-hour shifts (day/night) in continuous care services
* Being affiliated or entitled under a social security scheme
* Havinge received informed information about the study and have co-signed, with the investigator, a consent to participate in the study

Exclusion Criteria:

* Have made a tTrans meridian journey in the last month prior to the study
* Have a mMedically diagnosed sleep disorder such asof the hypersomnia or insomnia type
* Have a diagnosed and treated mental pathology
* Usually take a nap in the workplace in a quiet room
* Be pregnant or breastfeeding
* Have medically diagnosed neurovascular or neuromuscular pathologies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Evolution of reactive hyperemia index (RHI) | Change between week 1 and 12
  RHI is measured through the EndoPAT device® initially and at 12 weeks, and corresponds to the vascular reactivity following a 5-min occlusion on an arm

SECONDARY OUTCOMES:
Evolution of pulse wave velocity (PWV) | Change between week 1 and 12
  PWV is measured through the Popmeter® initially and at 12 weeks, and corresponds to the finger-o-foot pulse wave velocity(m/s)
Evolution of blood pressure | Change between week 1 and 12
  Systolic and diastolic blood pressure (mm Hg) measured in the sitting position in triplicate with an automatic blood pressure device (Panasonic EW3109) on the left arm, initially and at 12 weeks.
Evolution of heart rate variability (HRV) | Change between week 1 and 12
  24-h Holter-Electrocardiogram to derive temporal (SDNN, rMSSD, pNN50) and frequency (LF, HF, LF/HF) HRV indices initially and at 12 weeks.
Evolution of pro-inflammatory biomarkers | Change between week 1 and 12
  Fasting blood sample to measure hsCRP, IL-6 TNF-α, IL-1β initially and at 12 weeks.
Evolution of blood markers of endothelial function | Change between week 1 and 12
  Fasting blood sample to measure NO, SOD, IL-18 initially and at 12 weeks.
Evolution of subjective Fatigue | Change between week 1 and 12
  The Pichot fatigue scale (composed of 8 items, a score above 22 indicates excessive fatigue), initially and at 12 weeks.
Evolution of recovery Needs | Change between week 1 and 12
  French version of the Recovery Needs Scale (BRD), initially and at 12 weeks, wich consists of 11 items coded 0 or 1. A score is calculated for each participant, multiplied by 10 to give a score ranging from 0 to 100. The greater the need for recovery, the higher the score.
Evolution of state of health | Change between week 1 and 12
  The SF-36 questionnaire is used to assess quality of life, initially and at 12 weeks. It comprises 8 sub-scores ranging from 0 (minimum quality of life) to 100 (maximum well-being).
Evolution of sleep quality | Change between week 1 and 12
  Pittsburgh Sleep Quality Index (PSQI), initially and at 12 weeks : 24-question sleep quality assessment scale, a score > 5 indicates poor sleep quality.
Evolution of subjective sleepiness | Change between week 1 and 12
  Epworth questionnaire, initially and at 12 weeks : 8-question sleepiness assessment scale, a score above 10 indicates excessive sleepiness
Evolution of alertness at work assessed | Change between week 1 and 12
  The Karolinska Sleepiness Scale measures daytime sleepiness on a 9-point scale, based on 5 states and 4 intermediate states that are not verbally indicated, initially and at 12 weeks.
Evolution of sleep time | Change between week 1 and 12
  Actimeter measuring variations in wake-up and bedtimes, sleep duration, energy expenditure and time spent at different levels of physical activity intensity (sedentary, light intensity, moderate to intense intensity), initially and at 12 weeks.
Evolution of sleep duration | Change between week 1 and 12
  Actimeter measuring variations in wake-up and bedtimes, sleep duration, energy expenditure and time spent at different levels of physical activity intensity (sedentary, light intensity, moderate to intense intensity), initially and at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric ROCHE, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (1):
- Chu de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bouchou Y, Monnier M, Roche F, Pelissier C, Berger M. Effect of 12 weeks with a 30-min nap opportunity during the night shift of healthcare workers on early cardiovascular risk biomarkers: the NAPWORK study protocol of a randomised controlled trial. BMJ Open. 2026 Jan 22;16(1):e110108. doi: 10.1136/bmjopen-2025-110108. PMID 41571410